CLINICAL TRIAL: NCT05655364
Title: Development of a Breastfeeding Supportive Mobile Application: Examining the Effect of the Application on Breastfeeding Self-Efficacy and Outcomes in Primiparous
Brief Title: Development of a Breastfeeding Supportive Mobile Application
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Fatma Nilufer TOPKARA, Dr., Eskisehir Osmangazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: DBSMA
Record Dates: First submitted 2022-10-26; First posted 2022-12-19 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Breastfeeding; Self Efficacy; Postpartum
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental)
  Interventions: Other: Mobile application
- No intervention (No Intervention)

INTERVENTIONS:
Other: Mobile application — Breastfeeding Supportive Mobile Application
  Arms: Experimental

SUMMARY:
This work; The aim of this study was to develop a breastfeeding-supporting mobile application and to determine the effect of this application on breastfeeding self-efficacy and outcomes of primiparous. The research is planned to be carried out in two stages. In the first phase of the research, a mobile breastfeeding application based on Breastfeeding Self-Efficacy Theory will be developed. In the second phase of the study, a single-blind randomized pre-test-post-test control group intervention study design will be used to examine the effect of this developed application on breastfeeding self-efficacy and outcomes of primiparous.

The main questions it aims to answer are:

1. Does the breastfeeding-supporting mobile application based on the Breastfeeding-Self-Efficacy Theory change the breastfeeding-self-efficacy of women?
2. Does a breastfeeding support mobile application based on the Breastfeeding-Self-Efficacy Theory change the rate of women starting breastfeeding within the first hour after birth?
3. Does a breastfeeding-supporting mobile application based on the Breastfeeding-Self-Efficacy Theory change women's time to breastfeed alone?
4. Does a breastfeeding support mobile application based on the Breastfeeding-Self-Efficacy Theory change the breastfeeding duration of women?

DETAILED DESCRIPTION:
With the widespread adoption of smartphones and mobile software applications in healthcare delivery, developments in technology have significantly affected healthcare delivery models. Traditionally, only face-to-face interviews with health professionals have begun to be supported by mobile health applications (mHealth applications). An mHealth application refers to a standalone software application that can provide healthcare-related services through the use of portable devices such as smartphones. These applications provide more self-management in different health conditions and make it possible for individuals to access universal information, education and support network "anytime, anywhere" and therefore to receive care at home. Pregnant women and women who have just given birth are among the groups that most need and access health information online. They frequently use online applications to meet their need for information on birth and breastfeeding. In a systematic review of free-access mobile breastfeeding applications, it was revealed that there is a need to design a high-quality and interactive professional breastfeeding application that can encourage long-term breastfeeding behavior. It is thought that these practices have an important place in encouraging and supporting especially first-time mothers to breastfeed.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study,
* Being 18 years or older (18-45 years old),
* To know how to read and write in Turkish,
* Not having a visual-hearing disability,
* 24-36. to be between weeks of pregnancy,
* Being primiparous,
* Single pregnancy,
* Wanting to breastfeed,
* Not having received breastfeeding training in any period of pregnancy before,
* Using a smart phone,
* Absence of a diagnosed psychiatric illness.

Exclusion Criteria:

* Women carrying fetus with major anomaly,
* Women with breastfeeding contraindications,
* Women with high-risk pregnancies,
* Women who received advice from physicians not to breastfeed due to their health status, If the baby has any of the infectious or metabolic conditions specified by WHO or the Ministry of Health for which breastfeeding is contraindicated, When a baby with a birth weight of less than 2500 g is born or taken to the neonatal intensive care unit,
* When a baby with a birth weight over 2500 g is taken to the neonatal intensive care unit due to the week of birth, the mother will continue to receive information from the application, but will be excluded from the analysis.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2022-09-05 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Changing women's breastfeeding-self-efficacy | 8 months
  Changing women's breastfeeding-self-efficacy with a breastfeeding-supportive mobile application intervention based on the Breastfeeding-Self-Efficacy Theory
Changing the rate of women starting breastfeeding within the first hour after birth | 8 months
  Changing the rate of women starting breastfeeding within the first hour after birth with a breastfeeding-supportive mobile application intervention based on the Breastfeeding-Self-Efficacy Theory
Changing the duration of breastfeeding alone | 8 months
  Changing the duration of breastfeeding alone by women with a breastfeeding-supportive mobile application intervention based on the Breastfeeding-Self-Efficacy Theory
Changing the breastfeeding duration of women | 8 months
  Changing the breastfeeding duration of women with a breastfeeding-supportive mobile application intervention based on the Breastfeeding-Self-Efficacy Theory.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Nilüfer TOPKARA, Dr., Principal Investigator — Eskisehir Osmangazi University
Locations (1):
- Eskisehir Osmangazi University, Eskişehir, Turkey (Türkiye)